CLINICAL TRIAL: NCT06095739
Title: Study to Investigate the Effectiveness of a Topical Cosmetic Formulation DA-OTC-002
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Biology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AppliedBiology
Record Dates: First submitted 2023-10-11; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Hair Diseases; Alopecia; Hair Loss
MeSH Terms: conditions — Hair Diseases; Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DA-OTC-002 (Experimental): A 1mL topical application of DA-OTC-002 solution was applied to a 10cm x 10xm target area of the left side of the scalp of each subject.
  Interventions: Combination Product: DA-OTC-002

INTERVENTIONS:
Combination Product: DA-OTC-002 — The topical formula of DA-OTC-002 was formed from 2 molecules: an alpha 1 agonist (synephrine) and a TAAR receptor agonist
  A 1mL topical application of DA-OTC-002 was applied to a 10cm x 10xm target area of the right side of the scalp of each subject

SUMMARY:
The primary objective of the study was to assess the efficacy of DA-OTC-002 as a topical cosmetic hair treatment. The investigators conducted a prospective, institution-level, interventional, single-blinded, placebo-controlled investigation to assess the efficacy of a combination an alpha-1 agonist and a TAAR receptor agonist (DA-OTC-002) as a topical cosmetic hair treatment.

DETAILED DESCRIPTION:
76 female subjects were included in the study. Subjects were otherwise healthy females, aged 18 years are older, and had ample hair on the scalp to allow application of test article. Subjects with an interfering dermatologic disease or procedure, who were pregnant, lactating, or planning to become pregnant during the study, had experienced a clinically important medical event within 90 days of the visit, who were actively treated for hypertension, or had known allergies to any excipient in DA-OTC-002 were excluded from the study. This study was conducted in compliance with Good Clinical Practice, including the archival of essential documents. All subjects gave informed consent during the study enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Females Age 18 or older
* Willing and able to apply the treatment as directed, comply with study
* Subject has ample hair on the scalp to allow application of test article
* Otherwise healthy.
* Able to give informed consent

Exclusion Criteria:

* A medical history that may interfere with study objectives.
* Subjects with any dermatologic disease in the treatment area.
* Women who are pregnant, lactating, or planning to become pregnant during the study period.
* Subjects who have experienced a clinically important medical event within 90 days of the visit (e.g., stroke, myocardial infarction, etc).
* Subjects who are actively treated for hypertension.
* Subjects who have known allergies to any excipient in DA-OTC-002
* Subjects who are currently participating in another clinical study or have completed another clinical study with an investigational drug or device in the treatment area within 30 days prior to study treatment initiation.
* Subjects who have used any topical prescription medications in the treatment area within 30 days prior to study treatment initiation.
* Subjects who have had a dermatological procedure such as surgery in the treatment area within 30 days prior to study treatment initiation.
* Subject is unable to provide consent or make the allotted clinical visits.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2023-01-02 (Actual); Study Completion 2023-01-02 (Actual)

PRIMARY OUTCOMES:
Reduction in Hair Shedding Assessed by Target Area Hair Count Shedding | 30 minutes
  The average reduction in target area hair count after application of DA-OTC-002

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Fonesca, Principal Investigator — Applied Biology
Locations (1):
- Hospital Oscar Nicolau, Manaus, Brazil

IPD SHARING:
Plan to Share IPD: No